CLINICAL TRIAL: NCT04277039
Title: Effects of Osteopathic Treatment in Combination With Cognitive Training on Low Back Pain Patients: a Randomised Sham-controlled Trial
Brief Title: Effects of Osteopathic Treatment With Cognitive Training on Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Come Collaboration (Other)
Collaborators: Hospital General Universitario Santa Lucia (Other); Niguarda Hospital (Other); Orthoplus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COME-01-20
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
Keywords: osteopathic manipulative treatment; cognitive therapy; chronic low back pain; pain; disability
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Cognitive Training; Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OMT+CT (Experimental): It consists of 8 sessions of osteopathic treatment and two 20-min sessions of cognitive training per week per 2 months
  Interventions: Other: osteopathic treatment + cognitive training
- osteopathic treatment (Active Comparator): It consists of 8 sessions of osteopathic treatment throughout the 2-month study period
  Interventions: Other: osteopathic treatment
- usual care (Other): patients will continue the routine care as established by international guidelines
  Interventions: Other: usual care

INTERVENTIONS:
Other: osteopathic treatment + cognitive training — This intervention is a combination of manipulative osteopathic treatment and cognitive training to be administered each week for a 12-week study period
  Arms: OMT+CT
Other: osteopathic treatment — manual treatment using osteopathic procedure. 8 sessions for a 12 week study period
  Arms: osteopathic treatment
Other: usual care — administration of non-steroid inflammatory drug according to international guidelines
  Arms: usual care

SUMMARY:
The objective of this study is to verify whether the combined approach (osteopathic manipulative treatment -OMT- and cognitive training -CT) is more effective in the long term than the individual approaches (OMT or CT) in patients with chronic lumbar pain, evaluating the Numeric Rating Scale (NRS) and the Rolland-Morris Disability Questionnaire (RMDQ) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* aged between 30 and 65 y
* diagnosis of aspecific chronic low back pain
* minimum of 3 on the NRS score

Exclusion Criteria:

* Neuropathic pain or chronic widespread pain
* Low back spinal surgery in the last three years
* Low back spinal surgery to osteoporosis and/or traumatic fractures
* Rheumatic disease
* Pregnancy or having a baby in the last 12 months
* Painful disease in evidence through RX, MRI or CT in the last 6 months (listesis, moderate arthrosis, severe, algodystrophy etc.).
* The subjects have not to be treated with physical or manual therapies or psychotherapy in the last 6 months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in NRS at 3 months | 3 months
  Change from Baseline Numeric Rating Scale (NRS) of Pain at 3 months. NRS values range from 0-10, where 10 means highest pain and 0 no pain
Change in RMDQ at 3 months | 3 months
  Change from Baseline Rolland Morris Disability Questionnaire (RMDQ) at 3 months. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability)

SECONDARY OUTCOMES:
Changes in CSI | 1 month - 3 month - 6 month
  Baseline changes in Central Sensitization index (CSI). CSI values ranges from 0 to 100. A score of more than 40 indicates the presence of central sensitisation.
Changes in Oswestry | 1 month - 3 month - 6 month
  Baseline changes in Oswestry Low Back Pain Disability Questionnaire. The questionnaire range is from 0 to 100. Zero is equated with no disability and 100 is the maximum disability possible
BPQ | 1 month - 3 month - 6 month
  Baseline Changes in Body Perception Questionnaire
Changes in DASS-21 | 1 month - 3 month - 6 month
  Baseline changes in Depression Anxiety Stress Scales-21. The scale ranges from 0 to 36, where 36 indicates severe depression, anxiety and stress
Changes in SF-36 | 1 month - 3 month - 6 month
  Baseline changes in the Short Form-36. The questionnaire is a health survey ranging from 0 to 100. The lower the score the more disability.
Rate of AER | 1 month - 3 month - 6 month
  Number of participants with Adverse Events Reporting (AER) calculated by the rates
Changes in SCWT | 1 month - 3 month - 6 month
  Baseline changes in Stroop Color and Word Test. Word, color, and color-word T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal."
TMT | 1 month - 3 month - 6 month
  Trail Making Test
Change in NRS at 1 month | 1 month
  Change from Baseline Numeric Rating Scale (NRS) of Pain at 1 month. NRS values range from 0-10, where 10 means highest pain and 0 no pain
Change in NRS at 6 months | 6 months
  Change from Baseline Numeric Rating Scale (NRS) of Pain at 6 months. NRS values range from 0-10, where 10 means highest pain and 0 no pain
Change in RMDQ at 1 month | 1 month
  Change from Baseline Rolland Morris Disability Questionnaire (RMDQ) at 1 month. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability)
Change in RMDQ at 6 months | 6 months
  Change from Baseline Rolland Morris Disability Questionnaire (RMDQ) at 6 months. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cerritelli, PhD, Study Chair — Come Collaboration
Locations (3):
- Italy (3):
  - Santa Lucia Foundation, Rome, Lazio
  - Niguarda hospital, Milan, Lombardy
  - Orthoplus, Bolzano, Trentino-Alto Adige

IPD SHARING:
Plan to Share IPD: No
available upon request